CLINICAL TRIAL: NCT01110980
Title: Normalcy of Food Intake in Head and Neck Cancer Patients Receiving (Chemo)Radiotherapy Supported by Swallowing Therapy and Individual Dietary Counselling. (Supportive Care)
Brief Title: Normalcy of Food Intake in Head and Neck Cancer Patients
Acronym: FOCISD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Sorgente BV (Unknown); Fresenius Kabi Nederland BV (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FOCISD 01-03-2010
Record Dates: First submitted 2010-04-23; First posted 2010-04-27 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2012-10

CONDITIONS: Neoplasms, Head and Neck
Keywords: Head and Neck neoplasms; Radiotherapy; Diet counselling; Swallow therapy; Food intake
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Swallowing therapy (Experimental): Swallowing therapy in combination with individual dietary counselling
  Interventions: Other: Swallow therapy in combination with individual dietary counselling
- Individual dietary counselling (Active Comparator): Swallowing therapy only on indication. (usual care)
  Interventions: Other: Individual dietary counselling

INTERVENTIONS:
Other: Swallow therapy in combination with individual dietary counselling — Weekly swallowing therapy (by speech language therapist) from start of (chemo)radiation until 6 months after last (chemo)radiation. Weekly Individual dietary counselling (by dietician) form the start of (chemo) radiotherapy until 6 months after last (chemo)radiation. With close interaction between the both interventions.
  Other Names: PST+IDC
  Arms: Swallowing therapy
Other: Individual dietary counselling — Weekly Individual dietary counselling form the start of (chemo) radiotherapy until 6 months after last (chemo)radiation.
  Other Names: IDC
  Arms: Individual dietary counselling

SUMMARY:
* Background:

Oral nutrition appears to be a challenge for patients with head and neck cancer after radiotherapy. Many patients desire to (their) 'normal food intake' and return to oral nutrition with normal consistency without modifications and diet formulas. Due to the dysphagia experienced post treatment this seems tremendously difficult. Referral to a speech-language therapist for swallowing therapy is no standard procedure.

* Study design:

A prospective randomized study in patients with a tumor in Oral cavity, Nasopharynx, Oropharynx, Hypopharynx or Larynx with stage II-IV (UICC TNM-tumor classification), ≥ 18 years, eligible for primary treatment with (chemo)radiation or adjuvant radiotherapy with curative intent.

* Intervention:

Individually tailored swallowing therapy by an experienced speech-language therapist in cooperation with individual dietary counselling (by an experienced dietician, 'usual care') pre-, per- and post treatment (until 6 months after treatment). This might improve 'normalcy of food intake', quality (no food modifications) and quantity of food intake and besides decrease the use of tube feeding and/or nutritional supplements. Also patients quality of life and nutritional status may be influenced positively.

* Study hypothesis:

The purpose of this study is to determine whether combined individual swallowing therapy and individual dietary counselling in patients with head and neck cancer receiving (chemo)radiotherapy can improve 'normal food intake'. Food intake without modifications and tube feeding and/or nutritional supplements.

ELIGIBILITY:
Inclusion Criteria:

* Patients with tumor in oral cavity, nasopharynx, hypopharynx or larynx with stage II-IV (UICC TNM-tumor classification)
* Eligible for primary curative treatment intentions with (chemo)radiation or adjuvant (chemo)radiotherapy
* A signed informed consent

Exclusion Criteria:

* Historical swallowing problems (neurological or not tumor related)
* Unable to comprehend and carry out the swallowing rehabilitation
* Unable to answer study questions
* Radiation or surgery for head and neck cancer in history.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Normalcy of food intake | within 6 months
  Increase of "normalcy of food intake" of 10%

SECONDARY OUTCOMES:
Quality of life | within 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mattias A. W. Merkx, Prof. Dr., Study Director — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands